CLINICAL TRIAL: NCT00519363
Title: Statins and Lupus: Effects of Statins on Clinical Lupus Parameters, Serological Markers and Toll-like Receptors.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Center for Rheumatic Disease, Allergy, & Immunology (Other)
Collaborators: Saint Luke's Health System (Other)
Responsible Party: Nabih I Abdou, MD, PhD, Center for Rheumatic Disease Allergy & Immunology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-316; Saint; Luke's; Hospital; Grant
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; TLR's; Hyperlipidemia; age eighteen to sixty; female with SLE; SLEDAI, greater than four; LDL cholesterol elevated
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Hyperlipidemias; Hyperlipoproteinemia Type II | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 40mg, given orally daily for 3 months.
  Other Names: Lipitor 40mg

SUMMARY:
This is an open label pilot clinical trial on a cohort of 15 Lupus patients from the Center for Rheumatic Disease. Clinical evaluations and laboratory tests will be done and then if eligible, the patients will receive oral atorvastatin, at a fixed dose of 40mg/day. Statins have been shown to induce clinical improvement in rheumatoid arthritis patients, as well as lupus patients. The effectiveness has been noted within 8 to 14 days, we will do our study for 3 months. Clinical and laboratory tests will be checked at the 1 and 3 month interval. We hypothesize that statin drugs (atorvastatin) slow the progression of SLE(Systemic Lupus Erythematosus) disease activity and down regulates TLR(Toll-like receptors) 2,4,and 9 pathways in addition to lowering lipid levels.

DETAILED DESCRIPTION:
Atorvastin (Lipitor) is a commonly used drug approved by the FDA for treatment of dyslipidemias. It is a relatively safe drug to use with periodic monitoring.

Eligibility critera:

* age 18-60, females, as a marjority of lupus patients are female
* at least 4 ACR (American College of Rheumatology) criteria of SLE(Systemic Lupus Erythematosus)
* Moderate to Severe disease activity using approved SLEDAI(Systemic Lupus Erythematosus Disease Activity Index)
* LDL cholesterol 100-190mg/dl

Exclusion criteria:

* Pregnancy, and or lactating or wants to get pregnant
* Unable to take atorvastatin due to allergy, liver disease, elevated liver functions, myositis, or elvated CPK(creatine phosphakinase)
* already on lipid lowering therapy
* already on amiodarone, clarithromycin, cyclosporin, erythromycin, itraconazole, ketoconazole, nefazodone, verapamil, protease inhibitors, niacin, digoxin,k cholestyramine, colestipol
* has a dianosis of Myositis. Our goal is to colledt preliminary data to see if there is a trend for the efficacy of atorvastatin in ameliorating SLE disease activity and to evaluate TLRs(Toll-like receptor) in SLE patients. A p value of <0.05 will be considered statistically significant. Our baseline and at subsequent visits, we will have 80% power to detect a minimum of 34%-39% difference for most of the continous variables measured at different intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60, female
* have at least four ACR criteria for SLE
* SLEDAI score > 4
* LDL cholesterol level from 100-190mg/dl

Exclusion Criteria:

* Pregnant, lactating, or wanting to become pregnant
* unable to take atorvastatin due to allergy, liver disease, elevated lever function test, myositis, or eleveated CPK
* already on lipid lowering therapy
* participating in another lupus study
* on drugs such as: amiodarone, clarithromycin, clclosporine, erythromycin, itraconazole, ketoconazole, nefazodone, verapamil, protease inhibitors, niacin, digoxin, cholestryrmine, colestipol
* has a diagnosis of myositis

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
decrease the SLEDAI level of female lupus patients, down regulate the TLR 2,4, and 9. | 3 months

SECONDARY OUTCOMES:
lower lipid levels in female lupus patients | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nabih I Abdou, MD, PhD, Principal Investigator — The Center for Rheumatic Disease, Allergy, and Immunology
Locations (1):
- The Center for Rheumatic Disease, Allergy, and Immunology, Kansas City, Missouri, United States